CLINICAL TRIAL: NCT05569005
Title: A 3-year, 3-group, Preference, Multi-center Study to Demonstrate the Slowing of Disease Progression When Switching From Cigarette Smoking to the Tobacco Heating System (THS) in Mild to Moderate Chronic Obstructive Pulmonary Disease (COPD) Subjects With a History of Chronic Bronchitis Symptoms.
Brief Title: Effect of Switching From Cigarette Smoking to THS on Disease Progression in Mild to Moderate COPD Subjects With Chronic Bronchitis Symptoms.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study team decided to terminate the study due to operational infeasibility caused by challenges with recruiting the necessary number of participants.
Sponsor: Philip Morris Products S.A. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: P1-COPD-04-INT
Record Dates: First submitted 2022-09-30; First posted 2022-10-06 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: COPD; Smoking; Tobacco Use
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Smoking; Tobacco Use | interventions — Tobacco Products

STUDY DESIGN:
Intervention Model Description: A multiregional (Europe, U.S. and Asia) multi-center, open-label study with 3-group, parallel preference design (Cigarette, THS use and Smoking Abstinence).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- THS (Active Comparator): Subjects who are not willing to quit smoking.
  Interventions: Other: THS use
- Cigarette (Active Comparator): Subjects who are not willing to quit smoking.
  Interventions: Other: Cigarette
- Smoking Abstinence (Active Comparator): Subjects who are willing to quit smoking.
  Interventions: Other: Smoking Abstinence

INTERVENTIONS:
Other: THS use — Subjects who are not willing to quit smoking during the study duration will switch from cigarettes to using THS
  Other Names: Tobacco Heating System 3.0
  Arms: THS
Other: Cigarette — Subjects who are not willing to quit smoking during the study duration will continue smoking their own preferred brand of commercially available cigarettes.
  Arms: Cigarette
Other: Smoking Abstinence — Subjects who are willing to quit smoking may be prescribed an NRT to support them in remaining abstinent from use of any tobacco and nicotine containing products during the study. (Behavioral support will be provided to subjects to aid with abstinence.)
  Arms: Smoking Abstinence

SUMMARY:
The purpose of this study is to demonstrate the slowing of the disease progression including the improvement of Chronic Obstructive Pulmonary Disease (COPD) symptoms in smoking subjects with mild to moderate COPD and a history of chronic bronchitis symptoms (sputum and cough) who switch to the Tobacco Heating System (THS) as compared to those who continue to smoke cigarettes.

DETAILED DESCRIPTION:
This study will be a multiregional (Europe, U.S., and Asia) multi-center, open-label study with 3-group, parallel preference design (Cigarette, THS use, and Smoking Abstinence).

Subjects will self-select their group allocation according to their preference. Subjects who would like to quit cigarettes or THS during the study will be encouraged to do so and will be referred to appropriate services.

The study will be declared successful if a slowing of the disease progression is demonstrated with the primary objective endpoint of forced expiratory volume in the first second (FEV1) post-bronchodilator at Month 36 or if an improvement of COPD symptoms (COPD Assessment Test total score at interim analysis at Month 12) is demonstrated.

ELIGIBILITY:
Main Inclusion Criteria:

* Subjects have read, understood, and signed the written informed consent form (ICF)
* Diagnosis of COPD GOLD Stage 1 or 2 (FEV1/FVC <0.70 & FEV1 ≥60% predicted [post-BD])
* Current symptoms of chronic bronchitis (sputum and cough) based on CAT questionnaire scores for CAT1 (cough) item ≥ 3 and CAT2 (sputum) item ≥ 3
* Body mass index (BMI) 17.6-40.0 kg/m2 and body weight > 50 kg (male) or 40 kg (female).
* Subject has a smoking history of at least 10 years.
* Subject has been smoking ≥ 10 commercially available cigarettes/day on average (no brand restriction) for at least 1 year prior to V1 (based on self-reporting).
* Subject has not used other tobacco and nicotine products apart from cigarettes on a daily basis over the past year prior to V1.
* For subjects not willing to quit smoking only: have been advised to quit smoking, informed of smoking risks and of cessation programs and is still not willing to quit during the study duration.
* Subjects willing to quit smoking only: willing to set a target quit date (TQD) within the next 28 days at V1 as assessed by self-reported questions.

Main Exclusion Criteria:

* Subjects with any (mild, moderate or severe) COPD exacerbation that has not resolved at least four weeks prior to V1
* Subjects with active cancer or history of any cancer
* Subjects with pneumonia or other lower respiratory tract infections that have not resolved at least four weeks prior to V1
* Subjects with other active systemic infections that have not resolved at least 4 weeks prior to V1
* Subjects with other active respiratory disorders such as, but not limited to, tuberculosis, bronchiectasis, sarcoidosis, asthma2, pulmonary hypertension, interstitial lung diseases (e.g., idiopathic pulmonary fibrosis [IPF]). No new examination is required if the subject can present at V1, at a minimum, a Chest XRay (CXR) (or Computed Tomography (CT) of the chest, if available) not older than 6 months with anterior-posterior and left lateral views
* The subject is confirmed or suspected with active SARS-CoV-2 infection (as per site and per country recommendation)
* Clinically significant ECG alterations that will not allow subject to participate in the study, per Investigator's discretion
* Any concomitant disease that in the opinion of the investigator would interfere with the study procedures
* Subjects with diagnosed alpha-1 antitrypsin deficiency (AATD)
* History of alcohol and/or drug abuse which as per judgment of the Investigator would jeopardize either the participation in an investigational study or safety of the subject
* Positive serology test (HIV 1/2, hepatitis B or C).
* Inability to cooperate with the study procedures
* Previous participation in this study, or participation in an investigational study (drug or medical device) within 4 weeks before V1 (participation in observational studies/registries allowed)
* Close affiliation with the investigational site: a close relative of the investigator, a person dependent on the investigational site (e.g., employee or student of the investigational site)
* Subject is a current or former employee of the tobacco industry or their first-degree relatives (parent, child, spouse)
* Subjects have re-initiated smoking in the six months prior to V1
* Subjects have used in the past 3 months, or are currently daily using THS
* Any oral/injectable corticosteroids (acute or chronic treatments) or oxygen therapy in the last 2 months excluding short term use for a COPD exacerbation
* Female subject is pregnant or breastfeeding, (a urine pregnancy test will be performed at V1 and V2)
* For women of childbearing potential, female subject who does not agree to using an acceptable method of effective contraception during the entire study.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 715 (Actual)
Dates: Start 2022-12-16 (Actual); Primary Completion 2024-09-13 (Actual); Study Completion 2024-09-13 (Actual)

PRIMARY OUTCOMES:
Disease Progression | At month 36
  Disease progression will be assessed by measuring Forced Expiratory Volume in 1 second (FEV1), post-bronchodilator
COPD symptoms | At month 12
  COPD symptoms will be assessed from the total score of the COPD Assessment Test (CAT).

CONTACTS AND LOCATIONS:
Overall Officials: Christelle Haziza, PhD, Study Chair — Philip Morris Products S.A.
Locations (170):
- United States (81):
  - US49; Clinical Research of Brandon LLC, Brandon, Florida
  - US97; Riverside Research Group, Cape Coral, Florida
  - US38; Innovative Research Of West Florida, Inc., Clearwater, Florida
  - US47; Hope Clinical Trials, Inc, Coral Gables, Florida
  - UX24; Alfa Medical Research, Davie, Florida
  - US94; D & H Doral Research Center, LLC, Doral, Florida
  - UX10; Unique Clinical Trials, LLC, Doral, Florida
  - UX12; Solution Clinical Research, Doral, Florida
  - US83; Proactive Clinical Research LLC, Fort Lauderdale, Florida
  - UX01; 3Sync, Fort Lauderdale, Florida
  - US93; Finlay Medical Research, Greenacres City, Florida
  - US70; Harmony Medical Research Institute, Inc., Hialeah, Florida
  - US68; Global Research Associates, Homestead, Florida
  - US01; Accel Research Sites-LKD CRU, Lakeland, Florida
  - US25; Accel Research Sites, Largo, Florida
  - US12; Leesburg Medical Research Institute, LLC, Leesburg, Florida
  - US20; Accel Clinical Research, Maitland, Florida
  - UX15; Med-Care Research Corp., Miami, Florida
  - US13; LCC Medical Research Institute, LLC, Miami, Florida
  - US48; Ocean Clinical Research, LLC, Miami, Florida
  - US80; Enmanuel Advance Research Center, Miami, Florida
  - UX02; Finlay Medical Research, Miami, Florida
  - US84; Global Health Clinical Trials, Miami, Florida
  - US86; South Florida Research Center, Inc., Miami, Florida
  - US21; Bioclinical Research Alliance, Inc., Miami, Florida
  - US36; Allied Biomedical Research Institute, Miami, Florida
  - US79; Cordova Research Institute, LLC, Miami, Florida
  - US82; Florida International Medical Research, Miami, Florida
  - UX25; D&H National Research Centers (Bird), Miami, Florida
  - US72; BioMed Research and Medical Center. LLC, Miami, Florida
  - US55; American Research Institute, Miami, Florida
  - US56; Medical Research of Westchester, Inc, Miami, Florida
  - US95; Premier Research Associate, Inc, Miami, Florida
  - UX06; Wellness Research Center Inc, Miami, Florida
  - US37; Research Institute Of South Florida, Inc., Miami, Florida
  - US76; Reed Medical Research, Miami, Florida
  - US91; Ambert Medical Research, Miami, Florida
  - US90; Felicidad Medical Research, Miami, Florida
  - US40; Clinical Trials of Florida, LLC, Miami, Florida
  - UX07; Innovations Biotech, Miami, Florida
  - UX11; United Research Group, Miami, Florida
  - US43; San Marcus Research Clinic Inc, Miami Lakes, Florida
  - US89; 3Sync Research - Hialeah, Miami Lakes, Florida
  - US98; MedQuest Translational Sciences, Miami Lakes, Florida
  - UX26; Harmony Clinical Research, Inc, North Miami Beach, Florida
  - UX17; AES Orlando, Orlando, Florida
  - US04; Omega Research Consultants, Orlando, Florida
  - US10; Florida Institute for Clinical Research, Orlando, Florida
  - US57; Innovation Medical Group LLC, Palmetto Bay, Florida
  - US58; Bioresearch Institute LLC, Pembroke Pines, Florida
  - US41; Clinovation International Corp, Sebring, Florida
  - UX08; TBC Research Corp., Tamarac, Florida
  - US50; Precision Research Center, Tampa, Florida
  - UX04; Clinical Trials of Tampa, Tampa, Florida
  - US46; Palm Beach Research Center, West Palm Beach, Florida
  - US45; Clinical Site Partners, Inc. d/b/a CSP Orlando, Winter Park, Florida
  - US45; Clinical Site Partners, LLC - Winter Park, Florida Premier Research Institute (FPRI), Winter Park, Florida
  - UX99; Accelerated Enrollment Solutions (AES), Atlanta, Georgia
  - US81; Oracle Clinical Research, College Park, Georgia
  - UX22; ClinCept, LLC, Columbus, Georgia
  - US63; Lifeline Primary Care/CCT Research, Lilburn, Georgia
  - US31; IACTHealth d/b/a Centricity Research, Rincon, Georgia
  - US03; Inquest Clinical Research, Baytown, Texas
  - UX20; Novel Research, LLC, Bellaire, Texas
  - US42; Houston Pulmonary and Sleep Associates, Cypress, Texas
  - UX34; Mt.Olympus Medical Research, Friendswood, Texas
  - US88; HDH Research Inc, Houston, Texas
  - US73; Victorium Clinical Research, Houston, Texas
  - US53; Alpha Research Institute, LLC, Houston, Texas
  - US87; Biopharma Informatic Research Center, Houston, Texas
  - UX14; Prolato Clinical Research Center, Houston, Texas
  - UX09; Pioneer Research Solutions, Inc, Houston, Texas
  - UX18; Accurate Clinical Research, Inc, Humble, Texas
  - US39; Proactive Clinical Research, LLC (formerly Invesclinic, U.S. LLC), McAllen, Texas
  - US62; Metroplex Pulmonary And Sleep Medicine Center, McKinney, Texas
  - UX16; Pioneer Research Solutions, Inc, Mesquite, Texas
  - UX13; Synapse Clinical Research Inc., Missouri City, Texas
  - US59; Pulmonary and Sleep Institute, San Antonio, Texas
  - US52; Sherman Clinical Research, Sherman, Texas
  - UX21; R & H Clinical Research, Stafford, Texas
  - US74; Renovatio Clinical - The Woodlands Research Center, The Woodlands, Texas
- Bulgaria (26):
  - BG30; MHAT Puls AD, Blagoevgrad
  - BG28; MC Dr Staykov, Burgas
  - BG03; Medical Center Asklepii OOD, Dupnitsa
  - BG36; MHAT Sveti Ivan Rilski, Dupnitsa
  - BG05; Medical Center Pulmo-2018 EOOD, Haskovo
  - BG19; MC Zdrave 1, Kozloduy
  - BG17; Diagnostic Consultative Center 1 - Lom EOOD, Lom
  - BG07; Medical Center Leo Clinic, Lovech
  - BG26; Medical Center Hera - Montana branch, Montana
  - BG37; DCC (Diagnostic Consultative Center) 1 Pernik, Pernik
  - BG32; Medconsult Pleven, Pleven
  - BG40; Multiprofile Hospital for Active Treatment Trimontium, Plovdiv
  - BG12; MHAT Sveti Panteleymon EOOD, Plovdiv
  - BG08; Medical center Respiro, Razgrad
  - BG27; Diagnostic Consultative Center 1- Sliven EOOD, Sliven
  - BG29; MHAT Sliven to MMA Sofia, Sliven
  - BG33; Diagnostic Consultative Centre Sliven, Sliven
  - BG06; University First Multiprofile Hospital for Active treatment-Sofia EAD, Sofia
  - BG31; Medical Center Hera EOOD, Sofia
  - BG21; MC Preventsia 2000, Stara Zagora
  - BG38; MHAT Prof. Stoyan Kirkovich, Stara Zagora
  - BG01; Medical Center Zara EOOD, Stara Zagora
  - BG16; Medical Centre Leo Clinic EOOD, Varna
  - BG14; Medical Center Tara OOD, Veliko Tarnovo
  - BG39; Specialized Hospital for Active Treatment of Pneumo-phthizilogic Diseases - Dr. Treiman - Dr. Treiman, Veliko Tarnovo
  - BG22; SHATPPD Vratsa, Vratsa
- Czechia (13):
  - CZ05; Ordinace Hradebni s.r.o., České Budějovice
  - CZ09; Plicni ambulance Kralupy, s.r.o., Kralupy nad Vltavou
  - CZ07; MUDr. Jakub Strincl s.r.o., Liberec
  - CZ10; Nemocnice Mesice, Měšice
  - CZ17; Ordinace Pro Tbc a Respiracni Nemoci s.r.o, Olomouc
  - CZ06; PreventaMed, s.r.o., Olomouc
  - CZ02; Clinitrial, s.r.o., Prague
  - CZ16; Synexus Czech, s.r.o, Prague
  - CZ03; Praglandia s.r.o., Prague
  - CZ04; Zdravi-fit, s.r.o., Protivín
  - CZ08; Medison s.r.o., Přeštice
  - CZ12; Ordinace pro TBC a Respiracni Nemoci - Strakonice, Strakonice
  - CZ01; Progerint s.r.o., Vysoké Mýto
- Germany (17):
  - DE15; Emovis GmbH, Berlin
  - De10; Rcms, Berlin
  - DE21; Velocity Clinical Research Germany GmbH, Berlin
  - DE19; Synexus Clinical Research GmbH, Berlin
  - DE30; MECS Cottbus GmbH, Cottbus
  - DE28; Klifeck GmbH, Delitzsch
  - DE07; Klinische Forschung Dresden GmbH, Dresden
  - DE26; Synexus Clinical Research GmbH, Frankfurt
  - DE06; Klinische Forschung Hamburg GmbH, Hamburg
  - DE03; Klinische Forschung Hannover-Mitte GmbH, Hanover
  - DE01; Leipzig Research Centre-Synexus Clinical Research GmbH, Leipzig
  - DE04; Facharzt fur Innere Medizin und Pneumologie, Leipzig
  - DE12; Studienzentrum FMZ, Leipzig
  - DE17; Klinische Forschung Berlin-Mitte, Mitte
  - DE27; Centrum fuer Diagnostik und Gesundheit (CDG), Munich
  - DE25; Gemeinschaftspraxis Dres. Holger Kittner und Kerstin Hartig, Naunhof
  - DE14; Studienzentrum Dr.med.Schlenska, Peine
- Japan (12):
  - JP05; Tashiro Endocrinology Clinic, Fukuoka, Fukuoka
  - JP11; Haruta Respiratory Clinic, Hiroshima, Hiroshima
  - JP12; Takahashi Internal Medicine and Respiratory Clinic, Obihiro-shi, Hokkaido
  - JP14; Sawada Clinic, Himeji-Shi, Hyōgo
  - JP09; Takahashi Internal Medicine, Kawasaki, Kanagawa
  - JP08; Uchiyama Clinic, Jōetsu, Niigata
  - JP10; Yamagata Clinic (Goto-J Respiratory and Allergy Clinic), Ōita, Oita Prefecture
  - JP03; Tokyo-Eki Center, Chuo-Ku, Tokyo
  - JP01; Fukuwa Clinic, Chuo-Ku, Tokyo
  - JP02; P-one Clinic, Hachioji-shi, Tokyo
  - JP06; Higashi Shinjuku Clinic, Shinjuku-ku, Tokyo
  - JP04; Sanyudo Hospital, Yonezawa-shi, Yamagata
- Romania (3):
  - RO05; Centrul Medical de Diagnostic si Tratament Ambulatoriu Neomed SRL, Brasov
  - RO04; Sc Sana Monitoring Srl, Bucharest
  - RO06; Sc Ames Research Srl, Călăraşi
- Slovakia (11):
  - SK04; DIVERSITAS s.r.o. - Hlohovec vseobecne, Hlohovec
  - SK08; IRS - Medicínska cinnost s.r.o., Košice
  - SK01; PANACEUM s.r.o., Košice
  - SK02; MEDI M&M s.r.o., Moldava nad Bodvou
  - SK07; Hodosi-MED s.r.o., Moldava nad Bodvou
  - SK05; MEDIPA, s.r.o., Vseobecna ambulancia pre dospelych, Piešťany
  - SK12; PULMO s.r.o., Prešov
  - SK06; MUDr. Viliam Cibik, Phd, s.r.o., Pruské
  - SK10; Plucna ambulancia Hrebenar s.r.o., Spišská Nová Ves
  - SK09; Aquilamed s. r. o., Štiavnik
  - SK03; Alergia, s.r.o., Topoľčany
- United Kingdom (7):
  - GB07; Egin Research Ltd, High Wycombe, Buckinghamshire
  - GB05; Accellacare South London, Orpington, Kent
  - GB06; Velocity Clinical Research North London, North Finchley, London
  - GB04; Accellacare North London, Northwood, Middlesex
  - GB03; Accellacare Northamptonshire, Corby, Northamptonshire
  - GB02; Accellacare Warwickshire, Coventry, West Midlands
  - GB01; Accellacare Yorkshire, Shipley, Yorkshire